CLINICAL TRIAL: NCT00401817
Title: Phase II Study of Bevacizumab Plus CHOP-Rituximab in Patients With Untreated Mantle Cell Lymphoma (NHL)
Brief Title: Bevacizumab + CHOP-Rituximab in Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0604008463
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Untreated Mantle Cell Lymphoma
MeSH Terms: interventions — Bevacizumab; Rituximab

ARMS (1):
- Study Treatment Arm (Experimental): Bevacizumab-R-CHOP therapy included bevacizumab administered at 15 mg/kg on day 1, and standard dose R-CHOP on day 3, for six 21-day cycles
  Interventions: Drug: Bevacizumab; Drug: Rituximab; Drug: CHOP

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg on day 1 of each of 6 cycles
Drug: Rituximab — Rituximab will be administered prior to CHOP on day 3 of every cycle for a total of 6 cycles.
  The dose to be administered is:
  Rituximab: 375 mg/m2
Drug: CHOP — Standard CHOP chemotherapy will be administered at full dose every 21 days for a total of 6 cycles. The doses to be used are: Cyclophosphamide: 750 mg/m2 IV on day 3 Doxorubicin: 50 mg/m2 IV on day 3 Vincristine: 1.4 mg/m2 IV (not to exceed 2.0 mg total) on day 3 Prednisone: 100 mg PO days 3 - 7

SUMMARY:
Primary Objective

1. To evaluate the safety profile of Bevacizumab (Bevacizumab™)- Rituximab (Rituxan®)-CHOP (RA-CHOP) in patients with newly diagnosed mantle cell lymphoma (MCL).

Secondary Objectives

1. To evaluate the response rate and time to disease progression of the RA-CHOP regimen in patients with newly diagnosed MCL.
2. To prospectively characterize the angiogenic profiles of MCL patients during RA-CHOP treatment.

DETAILED DESCRIPTION:
Bevacizumab administered at 15 mg/kg on day 1 of each of 6 cycles

Rituximab administered 375 mg/m2 on day 3 of each of 6 cycles (with usual premedications)

Standard CHOP chemotherapy administered on day 3 every 21 days (full dose) for 6 cycles of treatment

Once completed six cycles of therapy (~18 weeks), patients will be evaluated every 3 months for the first year post treatment, then every 6 months until disease progression or death for years 2 through 5 post treatment. Patients who have disease progression will be contacted every 6 months until death to assess for survival status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of mantle cell Non-Hodgkin's Lymphoma with characteristic immunophenotypic profile: CD5(+), CD19(+) or CD20(+), cyclin D1(+), CD23(-) and CD10(-)
* Patient has not received any prior anti-cancer therapy for lymphoma
* Laboratory parameters (unless considered by investigator to be due to lymphoma):

Absolute neutrophil count > 1000 cells/mm3 Platelet count > 50,000 cells/mm3 Hemoglobin > 7 gm/dL Creatinine < 2.0 x ULN Total bilirubin < 2.0 x ULN

* Patient has at least one tumor mass > 1.5 cm in one dimension
* Available tumor tissue for correlative studies (rebiopsy to be performed if needed)
* Patient is > 18 years old
* Patient has KPS > 50%
* Patient has signed IRB-approved informed consent
* Patient agrees to use birth control for duration of study

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma
* Known hepatitis infection
* Known HIV positivity
* Known history of renal disease with proteinuria; urine protein:creatinine ratio ³1.0 at screening
* Uncontrolled hypertension: blood pressure of >150/100 mmHg at screening
* Unstable angina
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Patient has ejection fraction < 50%
* Patient is taking coumadin, or has known history of thrombosis within last 6 months
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 1
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Serious, non-healing wound, ulcer, or bone fracture
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patient is pregnant or nursing
* Patient is receiving other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Leonard, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Weill Medical College of Cornell University, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Treatment Arm
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 60 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicity
Description: Number of patients with reversible myelosuppression (Primary toxicity was reversible myelosuppression) Toxicities were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
Time Frame: 38 months
Measure: Number; unit: participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 11
participants | 8

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate measured using Kaplan-Meier survival analysis
  Response criteria were those reported by Cheson et al. (1999)
Time Frame: 38 Months (min 33 months, max 62 months)
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 11
percentage of participants | 82 [48 to 98]

3. Secondary Outcome: Progression-Free Survival
Description: The percentage of patients who have not progressed at the three year time point.
  The 3-year PFS rate was estimated based on the Kaplan-Meier analysis.
Time Frame: 3 years
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Study Treatment Arm: Bevacizumab-R-CHOP therapy included bevacizumab administered at 15 mg/kg on day 1, and standard dose R-CHOP on day 3, for six 21-day cycles
  Bevacizumab: 15 mg/kg on day 1 of each of 6 cycles
  Rituximab: Rituximab will be administered prior to CHOP on day 3 of every cycle for a total of 6 cycles.
  The dose to be administered is:
  Rituximab: 375 mg/m2
  CHOP: Standard CHOP chemotherapy will be administered at full dose every 21 days for a total of 6 cycles. The doses to be used are: Cyclophosphamide: 750 mg/m2 IV on day 3 Doxorubicin: 50 mg/m2 IV on day 3 Vincristine: 1.4 mg/m2 IV (not to exceed 2.0 mg total) on day 3 Prednisone: 100 mg PO days 3 - 7
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 11
percentage of patients | 23 [4 to 51]

4. Secondary Outcome: Overall Survival
Description: The percentage of patients who have survived at the three year time point.
  The 3-year OS rate was estimated based on the Kaplan-Meier analysis.
Time Frame: 3 years
Population: Evaluable Patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 11
percentage of patients | 82 [45 to 95]

ADVERSE EVENTS:
Arm/Group | Study Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Arm (N=11)
Prostate Cancer (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment Arm (N=11)
Neutropenia (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Febrile Neutropenia (Infections and infestations) | 1
Infection (normal ANC) (Infections and infestations) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Bleeding (General disorders) | 1
Rituximab infusion rxn (Infections and infestations) | 4
Neuropathy (Nervous system disorders) | 4
Fatigue (General disorders) | 7
Hypocalcemia (Blood and lymphatic system disorders) | 4
Constipation (General disorders) | 3
Edema (General disorders) | 3
Nausea (General disorders) | 2
Second malignancy (General disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Mouth sore (General disorders) | 2
Hyperkalemia (Blood and lymphatic system disorders) | 2
Hypoalbuminemia (Blood and lymphatic system disorders) | 2
Congestive heart failure (Cardiac disorders) | 1
Dyspnea (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes